CLINICAL TRIAL: NCT00648479
Title: New Method for Distal Interlocking of Cannulated Intramedullary Nails
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the company does not want to proceed yet with the study
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EKL-001-HMO-CTIL
Record Dates: First submitted 2008-03-17; First posted 2008-04-01 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Fracture
Keywords: Fracture Fixation
MeSH Terms: conditions — Fractures, Bone | interventions — Fluoroscopy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Device: The Guiding Star
- 2 (Active Comparator)
  Interventions: Device: fluoroscopy (OEC 9800 - General Electric)

INTERVENTIONS:
Device: The Guiding Star
  Arms: 1
Device: fluoroscopy (OEC 9800 - General Electric)
  Arms: 2

SUMMARY:
We intend to include10 patients in this study and trial. Prior to treatment they will sign an informed consent form, stating that they are acquainted with the surgical procedure and study, and that they consent to participate in the study.

Five patients will undergo regular operation with Universal tibial reamed nail (AO-Synthes) using the fluoroscopy device: OEC 9800 (GENERAL ELECTRIC). five patients will undergo the same operation using the new navigation system:"The Guiding star" method.

The allocation will be random.

ELIGIBILITY:
Inclusion Criteria:

1. Signing Informed consent.
2. Conscious patients.

Exclusion Criteria:

1. Hemodynamic Instability.
2. Multiple system injuries.
3. Pregnancy.
4. Soldiers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)

PRIMARY OUTCOMES:
the outcome will be asses using regular fluoroscopy in the operation room.